CLINICAL TRIAL: NCT01405300
Title: The Effects of Peanuts and Peanut Products on Glucose Control and Vascular Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Peanut Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PKE PPNUT
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peanut (Experimental)
  Interventions: Dietary Supplement: Peanut
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Control — 34.8 g dextrose, 150 g heavy whipping cream, 39g chocolate syrup, 15 g sunflower oil, 22 g safflower oil, 27 g powdered egg whites, 9.6 g of fiber supplement, water and crushed ice. It will deliver ~1200 kcal.
  Arms: Control
Dietary Supplement: Peanut — 34.8 g dextrose. 137 g heavy whipping cream, 39g chocolate syrup + 3 oz peanuts with skin. It will deliver ~1200 kcal.
  Arms: Peanut

SUMMARY:
Pilot study data have demonstrated that peanuts ameliorate the postprandial glucose and insulin response when incorporated into an acute high fat/high glucose meal. However, it is unclear whether acute consumption of peanuts can also influence vascular function. This study will therefore evaluate the effects of acute peanut consumption on vascular function, glycemic control, and plasma lipids. The hypothesis is that that addition of peanuts to a high fat/high glucose meal will reduce the production of triglycerides, glucose, and improve endothelial function as measured by flow-mediated dilation (FMD).

ELIGIBILITY:
Inclusion Criteria:

* 20-50 years of age
* LDL-C below 160 mg/dL
* Triglyceride below 350 mg/dL
* Blood pressure within normal ranges (below 140/90 mmHg)
* Not taking medication for elevated lipids, blood pressure or glucose

Exclusion Criteria:

* Allergies to peanuts or dairy products
* Known intolerance for high fat meals
* History of cardiovascular disease (CVD), kidney disease, diabetes or inflammatory diseases such as GI disorders and arthritis
* Use of non-steroidal anti-inflammatories or immunosuppressants
* Conditions requiring the use of steroids
* Use of medication or supplements for elevated lipids, blood pressure or glucose
* Donation of blood or plasma during the study
* History of thyroid disease
* Women
* Lactose intolerance

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Flow-Mediated Dilation at 4 hours postprandial | 0 min; 240 min

SECONDARY OUTCOMES:
Change from baseline in oxidative stress over 4 hours postprandial | 0 min, 30 min, 60 min, 120 min, 240 min
Change from baseline in serum lipids over 4 hours postprandial | 0 min, 30 min, 60 min, 120 min, 240 min
Change from baseline in serum glucose over 4 hours postprandial | 0 min, 30 min, 60 min, 120 min, 240 min
Change from baseline in serum insulin over 4 hours postprandial | 0 min, 30 min, 60 min, 120 min, 240 min

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, RD, Principal Investigator — Penn State University; Ann C Skulas-Ray, PhD, Study Director — Penn State University; Xiaoran Liu, Study Director — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Liu X, Hill AM, West SG, Gabauer RM, McCrea CE, Fleming JA, Kris-Etherton PM. Acute Peanut Consumption Alters Postprandial Lipids and Vascular Responses in Healthy Overweight or Obese Men. J Nutr. 2017 May;147(5):835-840. doi: 10.3945/jn.116.246785. Epub 2017 Mar 29. PMID 28356431